CLINICAL TRIAL: NCT06986148
Title: Comparing Antibiotic Treatment Strategies for Children With Community-Acquired Pneumonia in Outpatient Settings (Safety-Net Antibiotic Prescribing to Manage Pediatric Pneumonia [STAMPP])
Brief Title: Comparing Antibiotic Treatment Strategies for Children With Pneumonia in Outpatient Settings: (STAMPP)
Acronym: STAMPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Todd A. Florin, Associate Division Head for Academic Affairs & Research, Division of Emergency Medicine, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB_00185848; BPS-2023C3-35456 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2025-05-07; First posted 2025-05-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Community Acquired Pneumonia (CAP); Community Acquired Pneumonia
Keywords: Community-acquired Pneumonia; Pediatric Respiratory Diseases; Pneumonia; Antibiotic Use; SNAP
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Antibiotic Prescribing (Active Comparator): For participants randomized to this arm, a prescription is filled and the antibiotic is administered right after the index visit.
  Interventions: Other: Immediate Antibiotic Prescribing Group Instructions
- Safety Net Antibiotic Prescribing (SNAP) (Other): For participants randomized to this arm, a prescription is provided, but the patient is instructed not to take the antibiotic unless the child is not improving at 72 hours or sooner if getting worse.
  Interventions: Other: Safety Net Antibiotic Prescribing (SNAP) Group Instructions

INTERVENTIONS:
Other: Immediate Antibiotic Prescribing Group Instructions — Children randomized to the immediate antibiotic prescribing group will receive an antibiotic prescription with instructions to fill and administer the antibiotics.
  Arms: Immediate Antibiotic Prescribing
Other: Safety Net Antibiotic Prescribing (SNAP) Group Instructions — For children randomized to the SNAP group, their parents or guardians will receive a prescription for antibiotics, but will be told not to administer the antibiotic unless their child's symptoms show no improvement at 72 hours or worsen within 72 hours.
  Arms: Safety Net Antibiotic Prescribing (SNAP)

SUMMARY:
The goal of this clinical trial is to determine if a "watch and wait" antibiotic strategy, called Safety Net Antibiotic Prescribing (SNAP), can safely reduce unnecessary antibiotic use while ensuring that children diagnosed with community-acquired pneumonia get better from their illness. The main aims of this study are:

* To compare the effectiveness of SNAP versus immediate antibiotic prescribing in children with mild community-acquired pneumonia (CAP)
* To identify which patient groups benefit most from the SNAP strategy
* To identify factors that shape implementation of each prescribing strategy.

Researchers will compare the SNAP strategy (where parents or guardians are instructed to give antibiotics only if their child is not improving after 72 hours, or sooner if they are worsening) to the immediate antibiotic prescribing strategy (where parents or guardians are instructed to give the antibiotics right after their healthcare visit) to see if one strategy is more effective than the other.

Participants will be randomly assigned to either the immediate antibiotic group or the SNAP group at enrollment. Participation lasts 14 days with follow-up surveys at 4, 7, and 14 days after enrollment.

DETAILED DESCRIPTION:
This study is a multicenter, Hybrid Type-1effectiveness-implementation randomized clinical trial (RCT) designed to evaluate the effectiveness of a "Safety Net Antibiotic Prescribing" (SNAP) strategy versus an immediate antibiotic prescribing strategy for young children 12 months to <6 years of age with community-acquired pneumonia (CAP) who are treated as outpatients.

This study will recruit eligible patients from approximately 19 clinical sites consisting of pediatric emergency departments (EDs), primary care offices, and urgent care centers within the United States and enroll up to 2,000 patients. Patient recruitment will occur over a 3.5-year period. Participants will be identified and screened during routine visits at the clinical sites.

Through an online system, participants will be randomized to either the immediate antibiotic group or the SNAP group. All participants will receive a prescription for antibiotics as per usual care from their treating clinician.

The parents or guardians of the participants will be asked to complete an online survey on Days 4 and 14 (+/- 2 days) to collect data for the secondary outcomes, including quality of life, satisfaction, and return visits. On Day 7 (+/- 2 days), the parents or guardians of the participants will be contacted by phone to collect data for the primary outcome, focusing on clinical improvement and antibiotic use.

Acceptability and feasibility will be assessed with parent or guardian and clinician surveys and interviews. Parents or guardians will be surveyed at Day 14 and a subset will be invited for interviews within a month of the final follow-up visit. Clinicians will be surveyed, and a subset will be interviewed at the conclusion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Aims 1 and 2:
* Presenting with signs and symptoms of lower respiratory tract infection
* Diagnosed with community-acquired pneumonia (CAP) by a clinician
* The treating clinician intends to prescribe antibiotics for CAP, AND
* Well enough, as determined by the clinician at the time of the study enrollment visit, to be managed as an outpatient.
* Aim 3:
* Parent/guardian of child enrolled in the trial, OR
* Clinician who makes prescribing decision at the study site, OR
* Other practice-based parties (e.g. nurses, pharmacists, medical assistants, practice leaders) at study sites who can comment on the implementation of each prescribing strategy.

Exclusion Criteria:

* Aims 1 and 2:
* Hospitalization within the previous 7 days
* Oxygen saturation below 90%, if measured
* Incomplete immunization status (e.g., lacking at least 3 doses of the pneumococcal vaccines, typically given as part of the 2-, 4-, and 6-month vaccinations)
* Chronic medical conditions that increase the risk of bacterial CAP (e.g., chronic lung disease, cystic fibrosis, sickle cell disease),
* Substantially immunocompromised status (e.g., immunodeficiency, active cancer treatment, organ transplant with concurrent immunosuppressive agents)
* Receipt of oral or parenteral antibiotics within the previous 7 days
* Diagnosis of complicated pneumonia (e.g., empyema, lung abscess)
* Known bacterial source of infection warranting immediate antibiotics
* Pneumonia diagnosis within the previous 6 months, OR
* Prior enrollment in the trial
* Inability of the parent or guardian to speak English or Spanish
* Aim 3:
* Inability of the parent or guardian to speak English

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-07-16 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement | From enrollment to day 7
  Clinical improvement at 7 days after the index visit, defined as parent-reported (a) perception of overall improvement, (b) no worsening of fever, work of breathing, concerning changes in activity, or decreased oral intake, (c) no new antibiotic use or hospitalization following the index visit, and (d) improvement in at least one key pneumonia symptom in (b).
Antibiotic Use | From enrollment to day 7
  Antibiotic use through 7 days after the index visit, defined as Parent-reported antibiotic use (yes/no) at 7 days.

SECONDARY OUTCOMES:
Antibiotic Exposure | From enrollment to day 14
  Antibiotic exposure, defined as the number of days antibiotics were consumed through day 7 and day 14.
Clinical Improvement | From enrollment to day 14
  Clinical improvement at day 4 and day 14. Clinical improvement is defined as parent-reported perception of overall improvement, no worsening of fever, work of breathing, concerning changes in activity, or decreased oral intake, no new antibiotic use or hospitalization following the index visit, and improvement in at least one of these key pneumonia symptoms. Symptom improvement is assessed on an ordinal scale with "Much Worse" as the minimum measurement and "Much Better" as the maximum measurement.
Parent Satisfaction | From enrollment to day 14
  Parent-reported satisfaction with the treatment strategy at day 14. Parent-reported satisfaction with the treatment strategy is assessed on an ordinal scale with "Very Dissatisfied" as the minimum measurement and "Very Satisfied" as the maximum measurement.
Quality of Life Measures | From enrollment to day 14
  Quality of life, defined by parent/guardian using the Pediatric Quality of Life Inventory (PedsQL) at days 7 and 14
Return to Care | From enrollment to day 14
  Parent-reported return to medical care after index visit and reason for return

OTHER OUTCOMES:
Antibiotic-associated Adverse Events | From enrollment to day 14
  Rash, diarrhea, diaper dermatitis, oral thrush, vomiting, anaphylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Todd Florin, MD, MSCE, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Julia Szymczak, PhD, Principal Investigator — University of Utah
Locations (4):
- United States (4):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, a de-identified dataset will be prepared and made available for sharing with investigators as specified by the lead investigators and the funding agency. Data sharing will follow established guidelines to ensure that any shared dataset does not contain protected health information (PHI) and is fully anonymized. Investigators requesting access to the dataset will need to submit a data use agreement, specifying how the data will be used. Results of the study will be disseminated through peer-reviewed journals, presentations at scientific meetings, and the PCORI website.
  Aim 3 interview transcripts will not be shared to a publicly available repository since it will be impossible to fully anonymize the transcripts.